CLINICAL TRIAL: NCT05025592
Title: Conventional Transarterial Chemoembolization (cTACE) or Transarterial Chemoembolization (DEB-TACE) +HAIC Combined With Regorafenib ± Anti-PD1 Antibody for Unresected Hepatocellular Carcinoma
Brief Title: cTACE or DEB-TACE+HAIC Combined With Regorafenib ± Anti-PD1 Antibody for uHCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Zhu Xu, Hospital Chief Physician，MD, Peking University Cancer Hospital & Institute
Other Study IDs: 2021KT83
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: HCC; Transarterial Chemoembolization; Hepatic Arterial Infusion Chemotherapy; Regorafenib
MeSH Terms: interventions — regorafenib; spartalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- cTACE/DEB-TACE-HAIC+regorafenib±anti-PD1 antibody: patients will receive the combination treatment of cTACE/DEB-TACE plus HAIC and combined with regorafenib and anti-PD1 antibody or not. The anti-PD-1 antibody will be used depended on the contraindications or wishes of patients.
  Interventions: Drug: Regorafenib; Device: cTACE/DEB-TACE-HAIC

INTERVENTIONS:
Drug: Regorafenib — patients will received TACE-HAIC and regorafenib and anti-PD1 antibody or not
  Other Names: anti-PD1 antibody
Device: cTACE/DEB-TACE-HAIC — conventional transarterial chemoembolization(cTACE)/transarterial chemoembolization (DEB-TACE) plus hepatic artery infusion
  Other Names: conventional transarterial chemoembolization(cTACE)/transarterial chemoembolization (DEB-TACE) plus hepatic artery infusion

SUMMARY:
explore the effectiveness and safety of conventional transarterial chemoembolization (cTACE) or transarterial chemoembolization (DEB-TACE) plus hepatic arterial Infusion chemotherapy (HAIC) combined with regorafenib and anti-PD-1 antibody or not for unresected hepatocellular carcinoma (uHCC)

DETAILED DESCRIPTION:
This is a non-randomized, open, single-arm clinical study. Patients receive cTACE/DEB-TACE+HAIC treatment( 6-8 weeks as a cycle) and regorafenib and anti-PD1 antibody or not until the disease progresses, intolerable toxicity occurs, the patient is lost to follow-up or death, or situations other judged by researchers which treatment should be stopped.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate and sign the informed consent in writing;
2. Age: 18-75 years old;
3. No gender limit;
4. Unresectable hepatocellular carcinoma with clear pathological diagnosis or clinical diagnosis;
5. Unresectable hepatocellular carcinoma patients who failed first-line treatment (including but not limited to sorafenib, lenvatinib, atezolizumab combined with bevacizumab, etc.);
6. At least one measurable lesion (according to mRECIST criteria) imaging diagnosis time ≤ 21 days from selection;
7. Child-pugh grade A-B7 grade
8. The expected survival period is ≥3 months;
9. General physical condition (ECOG) 0-2;
10. Sufficient bone marrow hematopoietic function (within 7 days): hemoglobin ≥9 g/dL, white blood cells ≥3.0×10^9/L, neutrophils ≥1.5x 10^9/L, platelets ≥80x 10^9/L; liver and kidney functions are normal; (Within 14 days): TBIL≤1.5 times the upper limit of normal; ALT and AST≤5 times the upper limit of normal; creatinine≤1.5 times the upper limit of normal; INR≤1.7 or prolonged PT≤4s.

Exclusion Criteria:

1. Those who are currently receiving other effective treatments;
2. Patients who have received regorafenib in the past;
3. Patients who have participated in other clinical trials within 4 weeks before enrollment;
4. Unable to cooperate with cTACE and HAIC treatment;
5. Patients with primary malignant tumors other than hepatocellular carcinoma at the same time, except for cured skin basal cell carcinoma and cervical carcinoma in situ;
6. Clinically significant cardiovascular diseases, such as heart failure (NYHA III-IV), uncontrolled coronary heart disease, cardiomyopathy, arrhythmia, uncontrolled hypertension or a history of myocardial infarction within the past 1 year;
7. Neurological or mental abnormalities that affect cognitive ability, including central nervous system transfer;
8. There were active serious clinical infections (>grade 2 NCI-CTCAE version 4.0), including active tuberculosis within 14 days before enrollment;
9. Known or self-reported HIV infection;
10. Uncontrolled systemic diseases, such as poorly controlled diabetes;
11. Known to have hypersensitivity or allergic reactions to any component of the study drug;
12. Pregnancy (determined by serum β-chorionic gonadotropin test) or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with unresectable hepatocellular carcinoma are fail for fisrt line treatment((including but not limited to sorafenib, levatinib, atelizumab combined with bevacizumab, etc.) and will received cTACE/DEB-TACE plus HAIC and regorafenib and anti-PD1 antibody or not.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-10 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | 6 months
  The objective response rate (ORR) was defined as the complete response (CR) rate + the partial response (PR) rate
Progression free overall survival，PFS | 12 months
  PFS was defined as the interval between the time at which treatment was initiated and intrahepatic tumor and/or extrahepatic tumor progression, symptomatic progression, including massive ascites and liver function that was categorized as Child-Pugh grade C, or death from any cause
Overall survival，OS | 24 months
  overall survival (OS) was defined as the interval between the time at which treatment was initiated and death or the last follow-up assessment

SECONDARY OUTCOMES:
Disease control rate, DCR | 6 months
  disease control rate (DCR) was defined as the CR rate + the PR rate + the stable disease (SD) rate